CLINICAL TRIAL: NCT07311473
Title: Comprehensive Evaluation of Treatment Outcomes in Patients Treated With Palatal Temporary Skeletal Anchorage Devices
Brief Title: Comprehensive Outcomes of Palatal TSADs Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital of the Ministry of Interior, Kielce, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/2025/2
Record Dates: First submitted 2025-11-24; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Malocclusions
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palatal Temporary Skeletal Anchorage Devices (Experimental)
  Interventions: Device: Palatal temporary skeletal anchorage devices

INTERVENTIONS:
Device: Palatal temporary skeletal anchorage devices — Participants will receive orthodontic treatment involving the placement of palatal TSADs. Prior to the procedure, a cone-beam computed tomography (CBCT) scan will be obtained. Local anesthesia (0.2-0.5 mL) will be administered, after which two 2-mm diameter mini-implants will be inserted using a patient-specific surgical guide, and a palatal appliance will be positioned.

SUMMARY:
This study aims to evaluate clinical outcomes, patient-reported quality of life, the precision of surgical guides used for placing orthodontic mini-screws, and potential complications associated with the use of palatal temporary skeletal anchorage devices (TSADs) in orthodontically treated patients. The main questions it aims to answer are:

* What is the clinical effectiveness of palatal TSADs in orthodontic treatment outcomes?
* How do palatal TSADs affect the quality of life in orthodontic patients?
* How accurately do surgical guides transfer the digitally planned positions of mini-screws to their actual positions?
* What are the complications associated with the use of palatal TSADs in orthodontic treatment?

Participants will:

* Receive orthodontic treatment involving the placement of palatal TSADs
* Complete validated, standardized questionnaires assessing quality of life
* Be evaluated for skeletal and dental changes and monitored for clinical and technical complications throughout the course of treatment

ELIGIBILITY:
Inclusion Criteria:

* Presence of a malocclusion requiring palatal temporary skeletal anchorage devices (TSADs)
* No previous treatment involving TSADs
* Lack of systemic comorbidities
* Signed informed consent (and parental consent for minors)

Exclusion Criteria:

* Presence of uncontrolled systemic diseases or conditions that contraindicate orthodontic treatment or the placement of mini-screws
* Poor oral hygiene
* Allergies to materials used in mini-screws or associated orthodontic appliances
* Lack of patient consent for study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Change in maxillary width before and after TSAD-supported orthodontic treatment | Baseline (pre-treatment) and through completion of orthodontic treatment (up to 24 months).
  This primary outcome measure assesses changes in palatal width (in millimeters) among patients undergoing orthodontic treatment with temporary skeletal anchorage devices (TSADs). Measurements of palatal width will be conducted at two distinct time points: at baseline (prior to initiation of orthodontic treatment) and upon completion of the treatment. Measurements will be conducted using imaging techniques.

SECONDARY OUTCOMES:
Incidence and Types of Complications Associated with Orthodontic Treatment Using Palatal TSADs | Periprocedural period and up to 8 weeks post TSAD insertion.
  This secondary outcome measure is designed to evaluate the number, frequency, and types of complications specifically associated with TSADs and the palatal appliance during the periprocedural period and up to 8 weeks following TSAD insertion. The analysis will consider both the quantitative occurrence and qualitative characteristics of these early complications, providing insight into the short-term safety and clinical tolerability of TSAD-supported orthodontic therapy.
Patient-Reported Quality of Life During TSAD-Supported Use of the Palatal Appliance | Baseline (Day 0, day of appliance placement) through 8 weeks post-insertion.
  This secondary outcome measure evaluates patient-reported quality of life during the adaptation period to the palatal appliance supported by TSADs. On the day of appliance placement, patients will receive a self-administered questionnaire designed to assess subjective experiences related to wearing the appliance. The questionnaire includes, among others, items addressing discomfort or pain, difficulties during the initial adaptation phase, speech disturbances, or eating challenges. Completed questionnaires will be collected by the investigator at the subsequent orthodontic follow-up visit. The analysis will provide insight into the overall impact of the TSAD-supported palatal appliance on daily functioning.
Accuracy of Patient-Specific Surgical Guides for Palatal Mini-Screw Placement | Periprocedural (Day 0, immediately after placement of mini-screws using the surgical guide).
  This secondary outcome measure evaluates the precision of surgical guides used for the placement of palatal mini-screws during orthodontic treatment. Accuracy will be assessed by comparing the digitally planned positions of the mini-screws with their actual positions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ortostrefa Orthodontic Clinic, Nowy Sącz, Poland